CLINICAL TRIAL: NCT03917446
Title: Prediction of Volume Responsiveness After Propofol Bolus Injection in the Intensive Care Unit (ICU) Patients.
Brief Title: Volume Responsiveness Assesment After Propofol.
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radosław Owczuk, Professor, Medical University of Gdansk
Other Study IDs: JS-1
Record Dates: First submitted 2019-01-09; First posted 2019-04-17 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Circulatory Failure; Fluid Volume Disorder; Critical Illness
MeSH Terms: conditions — Shock; Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Euvolaemic: Patients with stroke volume variation less than 8%
  Interventions: Drug: Propofol bolus
- Hypovolaemic: Patients with stroke volume variation greater than 13%
  Interventions: Drug: Propofol bolus

INTERVENTIONS:
Drug: Propofol bolus — Each patient gets propofol bolus in three doses. 0.25 mg/kg, 0.5 mg/kg and 1 mg/kg. After each dose patient's blood pressure, heart rate and haemodynamic values calibrated with PICCO device (cardiac output, cardiac index, stroke index, stroke volume, stroke volume variation, dPmax) are recorded in 15 seconds intervals for 10 minutes.

SUMMARY:
Patients in ICU who suffer from circulatory insufficiency, regardless the cause that require invasive hemodynamic monitoring. The aim of the study is to correlate stroke volume variation which predicts fluid responsiveness with change of the blood pressure after intravenous admission of propofol. This test could become a surrogate of stroke volume variation in patients with contraindications to minimally invasive hemodynamic monitoring.

DETAILED DESCRIPTION:
This prospective, observational study was conducted after approval of the Independent Bioethics Commitee at Medical University of Gdańsk (numer zgody) and registered in ClinicalTrials.gov. Mechanically ventilated patients of intensive care unit who routinely recieved haemodynamic monitoring with PiCCO™ (Getinge AB, Sweden) technology using Philips IntelliVue PiCCO-Module (Philips Healthcare, Amsterdam, Netherlands), were enrolled. Patients were sedated with midazolam infusion at 0,15 to 0,6 mg kg-1 h-1 . Before the trial in each patient, heart rate (HR) invasive (IBP) and non - invasive blood pressure, (NIBP) infusion rate of catecholamines and non adrenergic vasopressors was recorded and PiCCO device was callibrated by transpulmonary thermodilution with 20 ml of cold saline. Global end diastolic volume (GEDV), intrathoracic blood volume (ITBV) and stroke volume variation (SVV) were calculated and recorded. For effective ventilation with increased tidal volume of 8 ml kg-1 of Predicted Body Weight, each patient recieved propofol bolus of 0,25 mg kg-1, 0,5 mg kg-1 and 1,0 mg kg-1 consecutively. Higher doses were used at good tolerance of the lower ones. After each bolus systolic and diastolic invasive blood pressure, heart rate (HR), continuous cardiac output (CCO), continuous cardiac index (CCI), stroke volume index (SI), stroke volume variantion (SVV), and left ventricular contractility index (dPmax) were recorded every fifteen seconds for ten minutes. The absolute and realtive change in blood pressure, compared to the values of blood pressure before the drug administration, were correlated with SVV. Time interval between each examination ranged from 4 to 48 hours.

ELIGIBILITY:
Inclusion Criteria:

ICU patient Haemodynamically instable Mechanically ventilated

Exclusion Criteria:

Simultaneous propofol infusion Contraindications for propofol Atrial fibrillation Valvular malfunction Aortic stenosis Aortic aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated ICU patients with heamodynamic instability aged above 18.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 10 minutes
  Change in blood pressure values after propofol bolus.
Heart rate | 10 minutes
  Change in heart rate values after propofol bolus.
Cardiac output | 10 minutes
  Change in cardiac output values after propofol bolus.
Cardiac index | 10 minutes
  Change in cardiac index values after propofol bolus.
Stroke volume | 10 minutes
  Change in stroke volume values after propofol bolus.
Stroke index | 10 minutes
  Change in stroke index values after propofol bolus.
Stroke volume variation | 10 minutes
  Change in stroke volume variation values after propofol bolus.
Maximum left ventricular contractility (dPmax) | 10 minutes
  Change in dPmax values after propofol bolus.

CONTACTS AND LOCATIONS:
Overall Officials: Jan J Stefaniak, M.D., Principal Investigator — Medical University of Gdansk, Faculty of Medicine
Locations (1):
- Medical University of Gdańsk - Departament of Anesthesiology and Intensive Care, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No